CLINICAL TRIAL: NCT03113331
Title: 3D Cohort Study: The Integrated Research Network in Perinatology of Quebec and Eastern Ontario
Brief Title: The 3D Cohort Study (Design, Develop, Discover)
Acronym: 3D
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: St. Justine's Hospital (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, William Fraser, Professor, Université de Sherbrooke
Other Study IDs: CRI 88413
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy Outcome
Keywords: Intrauterine growth restriction; Preterm birth; Birth defect; Infant growth; Neurodevelopmental outcomes
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal: blood, urine, vaginal secretions, nails, cord blood, placenta, hair, saliva Infant: hair, meconium, blood, urine, saliva Father: Blood, urine, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The 3D Cohort Study (Design, Develop, Discover) was established to help bridge knowledge gaps about the links between various adverse exposures during pregnancy with birth outcomes and later health outcomes in children.

DETAILED DESCRIPTION:
The main objective of the 3D study is to create a large pregnancy and birth cohort, allowing for the assessment of the effects of combined prenatal exposure on both birth outcomes and longer-term infant and child health. The specific objectives are to:

1. Determine the effects of pre- and post-natal exposures to environmental contaminants, nutritional factors and psychosocial stress on pregnancy and neurodevelopmental outcomes;
2. Assess the contribution of social, genetic, epigenetic, nutritional and environmental factors to the etiology and outcomes of intrauterine growth restriction (IUGR) and preterm birth; and
3. Assess the effects of assisted reproductive technologies (ART) on indicators of epigenetic modifications, and the relationship between such epigenetic changes and infant neurodevelopmental, cardiovascular, and metabolic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in French or English

Exclusion Criteria:

* Current intravenous drug use
* Severe illnesses or life threatening conditions
* Multiple gestation pregnancies

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The 3D Cohort Study is structured around a triadic (mother-partner-child) framework. The cohort comprises 2366 women recruited in the first trimester of pregnancy (8-14 weeks) who were planning to deliver in a collaborating hospital in the province of Quebec. Women and their partners were recruited between May 25, 2010 and August 30, 2012 at one of nine study centres during routine first-trimester prenatal visits to study hospitals and infertility clinics.
Sampling Method: Non-Probability Sample
Enrollment: 2366 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Intrauterine growth restriction | At delivery
  Birth weight smaller than 10th percentile
Preterm birth | At delivery
  Delivery before 37 weeks of gestation
Neurodevelopment - Bayley | When infants are 2 years old
  Neurodevelopmental assessment of the infant. Test used : Bayley Scales of Infant and Toddler Development (BSID-III; cognitive scale and motor scale combined). This test was done on 1520 children.
Neurodevelopment - ABAS | When infants are 2 years old
  Neurodevelopmental assessment of the infant. Test used : Bayley Adaptive Behaviour Questionnaire (ABAS-II). This test was done on 1520 children.
Neurodevelopment - Sensory Profile | When infants are 2 years old
  Neurodevelopmental assessment of the infant. Test used : Sensory Profile questionnaire. This test was done on 1520 children.
Neurodevelopment - MacArthur-Bates | When infants are 2 years old
  Neurodevelopmental assessment of the infant. Test used : MacArthur Communicative Development Inventories (CDI; French, English, Spanish and/or Mandarin). This test was done on 1520 children.
Neurodevelopment - M-CHAT | When infants are 2 years old
  Neurodevelopmental assessment of the infant. Test used : Modified Checklist of Autism in Toddlers (M-CHAT). This test was done on 1520 children.

CONTACTS AND LOCATIONS:
Overall Officials: William D Fraser, Dr, Principal Investigator — Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Fraser WD, Shapiro GD, Audibert F, Dubois L, Pasquier JC, Julien P, Berard A, Muckle G, Trasler J, Tremblay RE, Abenhaim H, Welt M, Bedard MJ, Bissonnette F, Bujold E, Gagnon R, Michaud JL, Girard I, Moutquin JM, Marc I, Monnier P, Seguin JR, Luo ZC; 3D Study Group. 3D Cohort Study: The Integrated Research Network in Perinatology of Quebec and Eastern Ontario. Paediatr Perinat Epidemiol. 2016 Nov;30(6):623-632. doi: 10.1111/ppe.12320. Epub 2016 Oct 25. PMID 27781295
- [Result] Morisset AS, Dubois L, Colapinto CK, Luo ZC, Fraser WD. Prepregnancy Body Mass Index as a Significant Predictor of Total Gestational Weight Gain and Birth Weight. Can J Diet Pract Res. 2017 Jun 1;78(2):66-73. doi: 10.3148/cjdpr-2016-035. Epub 2017 Feb 1. PMID 28145732
- [Result] Balayla J, Sheehy O, Fraser WD, Seguin JR, Trasler J, Monnier P, MacLeod AA, Simard MN, Muckle G, Berard A; 3D-Study Research Group From the Integrated Research Network in Perinatology of Quebec and Eastern Ontario. Neurodevelopmental Outcomes After Assisted Reproductive Technologies. Obstet Gynecol. 2017 Feb;129(2):265-272. doi: 10.1097/AOG.0000000000001837. PMID 28079770
- [Result] Shapiro GD, Seguin JR, Muckle G, Monnier P, Fraser WD. Previous pregnancy outcomes and subsequent pregnancy anxiety in a Quebec prospective cohort. J Psychosom Obstet Gynaecol. 2017 Jun;38(2):121-132. doi: 10.1080/0167482X.2016.1271979. Epub 2017 Jan 12. PMID 28079434
- [Result] Lamarre V, Gilbert NL, Rousseau C, Gyorkos TW, Fraser WD. Seroconversion for cytomegalovirus infection in a cohort of pregnant women in Quebec, 2010-2013. Epidemiol Infect. 2016 Jun;144(8):1701-9. doi: 10.1017/S0950268815003167. Epub 2015 Dec 21. PMID 26686548
- [Result] Pamidi S, Marc I, Simoneau G, Lavigne L, Olha A, Benedetti A, Series F, Fraser W, Audibert F, Bujold E, Gagnon R, Schwartzman K, Kimoff RJ. Maternal sleep-disordered breathing and the risk of delivering small for gestational age infants: a prospective cohort study. Thorax. 2016 Aug;71(8):719-25. doi: 10.1136/thoraxjnl-2015-208038. Epub 2016 Apr 15. PMID 27084956
- [Result] Reboul Q, Delabaere A, Luo ZC, Nuyt AM, Wu Y, Chauleur C, Fraser W, Audibert F. Prediction of small-for-gestational-age neonate by third-trimester fetal biometry and impact of ultrasound-delivery interval. Ultrasound Obstet Gynecol. 2017 Mar;49(3):372-378. doi: 10.1002/uog.15959. PMID 27153518
- [Result] Bisson M, Croteau J, Guinhouya BC, Bujold E, Audibert F, Fraser WD, Marc I. Physical activity during pregnancy and infant's birth weight: results from the 3D Birth Cohort. BMJ Open Sport Exerc Med. 2017 Jun 19;3(1):e000242. doi: 10.1136/bmjsem-2017-000242. eCollection 2017. PMID 28761717
- [Result] Thebault-Dagher F, Herba CM, Seguin JR, Muckle G, Lupien SJ, Carmant L, Simard MN, Shapiro GD, Fraser WD, Lippe S. Age at first febrile seizure correlates with perinatal maternal emotional symptoms. Epilepsy Res. 2017 Sep;135:95-101. doi: 10.1016/j.eplepsyres.2017.06.001. Epub 2017 Jun 10. PMID 28651086
- [Result] Tabatabaei N, Auger N, Herba CM, Wei S, Allard C, Fink GD, Fraser WD. Maternal Vitamin D Insufficiency Early in Pregnancy Is Associated with Increased Risk of Preterm Birth in Ethnic Minority Women in Canada. J Nutr. 2017 Jun;147(6):1145-1151. doi: 10.3945/jn.116.241216. Epub 2017 Apr 19. PMID 28424259
- [Result] Du Q, Luo ZC, Nuyt AM, Audibert F, Julien P, Wei SQ, Zhang DL, Fraser W, Levy E. Vitamin A and E Nutritional Status in Relation to Leptin, Adiponectin, IGF-I and IGF-II in Early Life - a Birth Cohort Study. Sci Rep. 2018 Jan 8;8(1):100. doi: 10.1038/s41598-017-18531-3. PMID 29311590
- [Result] He H, Nuyt AM, Luo ZC, Audibert F, Dubois L, Wei SQ, Abenhaim HA, Bujold E, Marc I, Julien P, Fraser WD; 3D Study Group. Maternal Circulating Placental Growth Factor and Neonatal Metabolic Health Biomarkers in Small for Gestational Age Infants. Front Endocrinol (Lausanne). 2018 Apr 25;9:198. doi: 10.3389/fendo.2018.00198. eCollection 2018. PMID 29922227
- [Result] Tabatabaei N, Eren AM, Barreiro LB, Yotova V, Dumaine A, Allard C, Fraser WD. Vaginal microbiome in early pregnancy and subsequent risk of spontaneous preterm birth: a case-control study. BJOG. 2019 Feb;126(3):349-358. doi: 10.1111/1471-0528.15299. Epub 2018 Jun 27. PMID 29791775
- [Result] Dubois L, Diasparra M, Bedard B, Colapinto CK, Fontaine-Bisson B, Tremblay RE, Fraser WD. Adequacy of nutritional intake during pregnancy in relation to prepregnancy BMI: results from the 3D Cohort Study. Br J Nutr. 2018 Aug;120(3):335-344. doi: 10.1017/S0007114518001393. Epub 2018 Jun 7. PMID 29875026
- [Result] Dupont C, Castellanos-Ryan N, Seguin JR, Muckle G, Simard MN, Shapiro GD, Herba CM, Fraser WD, Lippe S. The Predictive Value of Head Circumference Growth during the First Year of Life on Early Child Traits. Sci Rep. 2018 Jun 29;8(1):9828. doi: 10.1038/s41598-018-28165-8. PMID 29959368
- [Result] Bisson M, Tremblay F, Pronovost E, Julien AS, Marc I. Accelerometry to measure physical activity in toddlers: Determination of wear time requirements for a reliable estimate of physical activity. J Sports Sci. 2019 Feb;37(3):298-305. doi: 10.1080/02640414.2018.1499391. Epub 2018 Jul 14. PMID 30009665
- [Result] Dong Y, Luo ZC, Nuyt AM, Audibert F, Wei SQ, Abenhaim HA, Bujold E, Julien P, Huang H, Levy E, Fraser WD; 3D Cohort Study Group. Large-for-Gestational-Age May Be Associated With Lower Fetal Insulin Sensitivity and beta-Cell Function Linked to Leptin. J Clin Endocrinol Metab. 2018 Oct 1;103(10):3837-3844. doi: 10.1210/jc.2018-00917. PMID 30032199
- [Result] Guinhouya BC, Bisson M, Dubois L, Series F, Kimoff JR, Fraser WD, Marc I. Body Weight Status and Sleep Disturbances During Pregnancy: Does Adherence to Gestational Weight Gain Guidelines Matter? J Womens Health (Larchmt). 2019 Apr;28(4):535-543. doi: 10.1089/jwh.2017.6892. Epub 2018 Aug 1. PMID 30067134
- [Result] Choufani S, Turinsky AL, Melamed N, Greenblatt E, Brudno M, Berard A, Fraser WD, Weksberg R, Trasler J, Monnier P; 3D cohort study group. Impact of assisted reproduction, infertility, sex and paternal factors on the placental DNA methylome. Hum Mol Genet. 2019 Feb 1;28(3):372-385. doi: 10.1093/hmg/ddy321. PMID 30239726
- [Derived] Dubois L, Diasparra M, Bedard B, Colapinto CK, Fontaine-Bisson B, Morisset AS, Tremblay RE, Fraser WD. Adequacy of nutritional intake from food and supplements in a cohort of pregnant women in Quebec, Canada: the 3D Cohort Study (Design, Develop, Discover). Am J Clin Nutr. 2017 Aug;106(2):541-548. doi: 10.3945/ajcn.117.155499. Epub 2017 Jun 14. PMID 28615265